CLINICAL TRIAL: NCT01055509
Title: Effectiveness of Cognitive Adaptation Training Applied to Cognitive Impairment in Schizophrenia - A Randomised Trial
Brief Title: Compensatory Strategies Applied to Cognitive Impairment in Schizophrenia
Acronym: CAT-Denmark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Birte Oestergaard, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNR-2008037-1
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Social Adjustment; Quality of life; Recurrence; Hospitalization
MeSH Terms: conditions — Schizophrenia; Social Adjustment; Recurrence | interventions — Acclimatization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Adaptation Training (Experimental): Cognitive adaptation training and treatment as usual
  Interventions: Behavioral: Cognitive Adaptation Training
- Treatment as ususal (No Intervention): Pharmacological treatment, weekly contact to professionals (often in patient's homes), psychoeducation, social skill training in groups and psychosocial intervention with relatives.

INTERVENTIONS:
Behavioral: Cognitive Adaptation Training — All patients receive treatment as usual. Additionally, patients in the intervention arm receives training concerning solving concrete problems related to the patient's daily life using tools such as schedules, schemes and signs. Additional the patient can receive SMS messages or instructions for the use of schedules in cell-phones to prompt for activities. The intervention is conducted in the patients homes every 14th day in a period of six months.
  Other Names: Memory disorders; Adaptation
  Arms: Cognitive Adaptation Training

SUMMARY:
The purpose of this study is to determine whether Cognitive Adaptation Training are effective in comparison with conventional treatment, focusing on social functions, symptoms, relapse, re-hospitalisation, and quality of life in outpatients with schizophrenia.

DETAILED DESCRIPTION:
It is estimated that approximately 80% of patients with schizophrenia have reduced cognitive functions, representing problems with attention, verbal memory, short-term memory and executive functions (1-3). These impairments might have an impact on the patients ability to complete rehabilitation programmes, apply learned strategies to social problems, develop work skills and manage daily life (4,5). The effect of Cognitive Adaptation Training has been tested as a psychosocial treatment including training of compensatory strategies in order to sequence patient's adaptive behaviour, showing promising results concerning improved social functions (6). There are however no solid evidence for these statements. The existing few studies investigating the effect of Cognitive Adaptation Training (6-8) are underpowered (small sample sizes) and have a lack of younger patients, which limits the conclusions that can be drawn from the results of the improvement. The present trial employs a prospective design of 26 weeks with a follow-up period of 9 months after inclusion. The study will enroll 164 consecutively recruited participants from three Danish out-patient teams for young adults with a first episode of psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia.
* More than one year from referral to the psychiatric clinic.
* Receive mental medication and continual psychosocial treatment.
* Participants who have signed informed consent.

Exclusion Criteria:

* Participants who don't understand or speak Danish.
* Participants who live at an institution or who are long-term hospitalized.
* Participants who are unwillingly to complete protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in Social functioning assessed by Global Assessment of Function test and Health of the Nation Outcome Scales item 9-12 concerning social problems. | Baseline, six month and nine month.
  The effect of intervention on primary outcome are invetigated as longitudinal data at six and nine month. The data are analysed using mixed models.

SECONDARY OUTCOMES:
Changes in Social Functioning using Camberwell Assessment of Need questionnaire. Symptoms using Positive and Negative Syndrome Scale. Quality of Life using Lehman Quality of Life Interview-brief version. Relapse and frequency of hospitalization. | Baseline, six month and nine month.
  The effect of intervention on secondary outcome are invetigated as longitudinal data at six and nine month. The data are analysed using mixed models. However, relapse are analysed using survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lise Hounsgaard, PhD, Principal Investigator — Research Unit of Nursing
Locations (3):
- Denmark (3):
  - Early Intervention Team, Aabenraa
  - Schizophrenic Clinic, Psychiatric Department in Esbjerg and Ribe, Esbjerg N
  - Early Intervention Team, Odense

REFERENCES:
- [Background] Pfammatter M, Junghan UM, Brenner HD. Efficacy of psychological therapy in schizophrenia: conclusions from meta-analyses. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S64-80. doi: 10.1093/schbul/sbl030. Epub 2006 Aug 11. PMID 16905634
- [Background] Johnson-Selfridge M, Zalewski C. Moderator variables of executive functioning in schizophrenia: meta-analytic findings. Schizophr Bull. 2001;27(2):305-16. doi: 10.1093/oxfordjournals.schbul.a006876. PMID 11354597
- [Background] Kurtz MM, Moberg PJ, Ragland JD, Gur RC, Gur RE. Symptoms versus neurocognitive test performance as predictors of psychosocial status in schizophrenia: a 1- and 4-year prospective study. Schizophr Bull. 2005 Jan;31(1):167-74. doi: 10.1093/schbul/sbi004. Epub 2005 Feb 16. PMID 15888434
- [Background] Green MF, Kern RS, Braff DL, Mintz J. Neurocognitive deficits and functional outcome in schizophrenia: are we measuring the "right stuff"? Schizophr Bull. 2000;26(1):119-36. doi: 10.1093/oxfordjournals.schbul.a033430. PMID 10755673
- [Background] Brekke JS, Hoe M, Long J, Green MF. How neurocognition and social cognition influence functional change during community-based psychosocial rehabilitation for individuals with schizophrenia. Schizophr Bull. 2007 Sep;33(5):1247-56. doi: 10.1093/schbul/sbl072. Epub 2007 Jan 25. PMID 17255120
- [Background] Velligan DI, Diamond PM, Mintz J, Maples N, Li X, Zeber J, Ereshefsky L, Lam YW, Castillo D, Miller AL. The use of individually tailored environmental supports to improve medication adherence and outcomes in schizophrenia. Schizophr Bull. 2008 May;34(3):483-93. doi: 10.1093/schbul/sbm111. Epub 2007 Oct 10. PMID 17932089
- [Background] Velligan DI, Prihoda TJ, Ritch JL, Maples N, Bow-Thomas CC, Dassori A. A randomized single-blind pilot study of compensatory strategies in schizophrenia outpatients. Schizophr Bull. 2002;28(2):283-92. doi: 10.1093/oxfordjournals.schbul.a006938. PMID 12693434
- [Background] Velligan DI, Bow-Thomas CC, Huntzinger C, Ritch J, Ledbetter N, Prihoda TJ, Miller AL. Randomized controlled trial of the use of compensatory strategies to enhance adaptive functioning in outpatients with schizophrenia. Am J Psychiatry. 2000 Aug;157(8):1317-23. doi: 10.1176/appi.ajp.157.8.1317. PMID 10910797